CLINICAL TRIAL: NCT03324984
Title: Comparison of 1% Chloroprocaine vs. Hyperbaric Bupivacaine Spinals in Patients Undergoing Hemorrhoidectomies in an Ambulatory Surgery Center: A Double-Blind Randomized Controlled Pilot Trial.
Brief Title: 1% Chloroprocaine(PF) vs. Bupivacaine Spinals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-8414
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Return of Motor and Sensory Blockade; Anesthesia, Spinal; Decrease Discharge Time Status Post Hemorrhoidectomy
Keywords: Spinal anesthesia; Pain; Chloroprocaine
MeSH Terms: conditions — Pain | interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients, the researcher who recruited the patients and collected the data, nurse anesthetists, discharge anesthesiologist, and the Post Anesthesia Care Unit (PACU) nurse were all blinded to the patient treatment allocations. The operating room anesthesiologist (separate from the discharge anesthesiologist) was unblinded after receiving an enclosed envelope with the name of the spinal local anesthetic to perform the neuraxial anesthesia intraoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1% Chloroprocaine (PF) (Experimental): 1% Chloroprocaine is an ester-linked local anesthetic with the shortest duration of action of all local anesthetics.
  Interventions: Drug: 1% chloroprocaine
- 0.75% bupivacaine (Active Comparator): 0.75% bupivacaine is a amino-amide anesthetic local anesthetic. It is hyperbaric in nature due to addition of dextrose.
  Interventions: Drug: 0.75% bupivacaine

INTERVENTIONS:
Drug: 1% chloroprocaine — In 2018, 1% Chloroprocaine was approved by the FDA for spinal anesthesia use.
  Arms: 1% Chloroprocaine (PF)
Drug: 0.75% bupivacaine — Bupivacaine is used on label
  Arms: 0.75% bupivacaine

SUMMARY:
The use of 1% Chloroprocaine (PF) spinal anesthesia will reduce the recovery times and discharge time of patients undergoing hemorrhoidectomies as compared to 0.75% bupivacaine spinal. The primary objective is to compare the recovery times (return of motor and sensory function) and discharge time (voiding time) between 2-Chloroprocaine and 0.75% bupivacaine spinal anesthesia for hemorrhoidectomies. This is a randomized, prospective study assigning patients to either 2-Chloroprocaine (PF) or 0.75% bupivacaine spinal anesthesia group.

DETAILED DESCRIPTION:
The use of 1% Chloroprocaine (PF) spinal anesthesia will reduce the recovery times and discharge time of patients undergoing hemorrhoidectomies as compared to 0.75% bupivacaine spinal. The primary objective is to compare the recovery times (return of motor and sensory function) and discharge time (voiding time) between 1% Chloroprocaine and 0.75% bupivacaine spinal anesthesia for hemorrhoidectomies. This is a randomized, prospective study assigning patients to either 1% Chloroprocaine (PF) or 0.75% bupivacaine spinal anesthesia group. Consents for participation in the study will be obtained during the patients' preoperative anesthesia evaluation. There will be no change in the primary anesthetic technique (spinal anesthesia), since these patients routinely get spinal anesthesia for hemorrhoidectomies, however there would be a change in type of local anesthetic administration. On the day of surgery, consented patients will be randomized to one of the two groups. Both the patients and the researcher who recruited the patients and collected the data will be blinded. (Research assistant will hand an enclosed envelop to the anesthesiologists performing the spinal anesthesia with the name of local anesthetic to use) Postoperatively, the PACU nurse will be ask to document return of motor and sensory function in addition to voiding time. At the time of voiding, the nurse will be asked to inform an anesthesiologist (not involved in the case) for a postoperative evaluation and a discharge note. However, if the patient cannot void once there are able to ambulate, then they stay in PACU until they are the last patient in the unit. If still unable to void, the surgeon will be informed and an ultrasound bladder scan will be used to determine the volume of urine and the patient will be straight cath. The patient will be sent home and informed if he or she cannot void by the next day, then they should call the surgeon's office to notify them and go to the emergency room.

For postoperative data collection, the routine 24hr postoperative phone calls in which nurses make to patients will be utilize, however two additional questions will be asked, 1. Presence of nerve pain in the buttocks and thighs shooting down their legs unilaterally or bilaterally, 2. Inability to void, pass flatus or defecate. If any of the symptoms are present, then the nurse will inform an anesthesiologist (not involved in the case) whom will give the patient a call and advise them on treatment protocol. The research assistant will then be informed by the anesthesiologist who made the phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing anorectal procedures
* Age 18 and above
* American Society of Anesthesiologist Physical Status (ASA), I-III

Exclusion Criteria:

* Patient refusal
* Inability to understand and sign informed consent
* Allergic reaction to bupivacaine or other local anesthetics
* Coagulopathy (INR >= 1.5)
* Use of anticoagulant drugs (Plavix, Coumadin)
* Thrombocytopenia (Platelets < 100,000)
* Infection at the site
* Increased intracranial pressure
* Unstable spine, Spine abnormalities
* History of atypical cholinesterase (CP is metabolized by cholinesterase)
* Diagnosis of any disorders (i.e., benign prostatic hyperplasia, cystitis, vulvovaginitis) that would delay voiding
* Anticipated procedure time longer than 60 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elilary Montilla Medrano, MD, Principal Investigator — Montefiore Medicial Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfelbaum JL, Walawander CA, Grasela TH, Wise P, McLeskey C, Roizen MF, Wetchler BV, Korttila K. Eliminating intensive postoperative care in same-day surgery patients using short-acting anesthetics. Anesthesiology. 2002 Jul;97(1):66-74. doi: 10.1097/00000542-200207000-00010. PMID 12131105
- [Background] Liu SS, Strodtbeck WM, Richman JM, Wu CL. A comparison of regional versus general anesthesia for ambulatory anesthesia: a meta-analysis of randomized controlled trials. Anesth Analg. 2005 Dec;101(6):1634-1642. doi: 10.1213/01.ANE.0000180829.70036.4F. PMID 16301234
- [Background] Forster JG. Short-acting spinal anesthesia in the ambulatory setting. Curr Opin Anaesthesiol. 2014 Dec;27(6):597-604. doi: 10.1097/ACO.0000000000000126. PMID 25211156
- [Background] Pollock JE. Transient neurologic symptoms: etiology, risk factors, and management. Reg Anesth Pain Med. 2002 Nov-Dec;27(6):581-6. doi: 10.1053/rapm.2002.36457. No abstract available. PMID 12430108
- [Background] Fanelli A, Ghisi D, Allegri M. Is spinal anaesthesia a suitable technique for ultra-short outpatient procedures? Acta Biomed. 2013 Jun 1;84(1):76-80. PMID 24189768
- [Background] Smith KN, Kopacz DJ, McDonald SB. Spinal 2-chloroprocaine: a dose-ranging study and the effect of added epinephrine. Anesth Analg. 2004 Jan;98(1):81-88. doi: 10.1213/01.ANE.0000093361.48458.6E. PMID 14693591
- [Background] Vath JS, Kopacz DJ. Spinal 2-chloroprocaine: the effect of added fentanyl. Anesth Analg. 2004 Jan;98(1):89-94. doi: 10.1213/01.ANE.0000093360.02058.ED. PMID 14693593
- [Background] Kouri ME, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with lidocaine in volunteers. Anesth Analg. 2004 Jan;98(1):75-80. doi: 10.1213/01.ANE.0000093228.61443.EE. PMID 14693590
- [Background] Yoos JR, Kopacz DJ. Spinal 2-chloroprocaine for surgery: an initial 10-month experience. Anesth Analg. 2005 Feb;100(2):553-558. doi: 10.1213/01.ANE.0000130397.38849.4A. PMID 15673893
- [Background] Hejtmanek MR, Pollock JE. Chloroprocaine for spinal anesthesia: a retrospective analysis. Acta Anaesthesiol Scand. 2011 Mar;55(3):267-72. doi: 10.1111/j.1399-6576.2010.02371.x. PMID 21288208
- [Background] Pavlin DJ, Pavlin EG, Fitzgibbon DR, Koerschgen ME, Plitt TM. Management of bladder function after outpatient surgery. Anesthesiology. 1999 Jul;91(1):42-50. doi: 10.1097/00000542-199907000-00010. PMID 10422927
- [Background] Mulroy MF. Outpatients do not need to void after short neuraxial blocks. Anesthesiology. 2009 Dec;111(6):1388; author reply 1389. doi: 10.1097/ALN.0b013e3181bfa8d3. No abstract available. PMID 19934900
- [Background] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878
- [Background] Teunkens A, Vermeulen K, Van Gerven E, Fieuws S, Van de Velde M, Rex S. Comparison of 2-Chloroprocaine, Bupivacaine, and Lidocaine for Spinal Anesthesia in Patients Undergoing Knee Arthroscopy in an Outpatient Setting: A Double-Blind Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):576-83. doi: 10.1097/AAP.0000000000000420. PMID 27281722
- [Result] Kim SW, Khandaker R, Muse IO, Pulverenti T, Goman M, Patel J, Yedlin A, Balikai CP, Levine R, Choice C, Montilla Medrano E. Comparison of 1% chloroprocaine hydrochloride versus hyperbaric bupivacaine spinal in patients undergoing anorectal surgery in an ambulatory surgery center: a double-blind randomized clinical trial. Reg Anesth Pain Med. 2024 Dec 31:rapm-2024-106130. doi: 10.1136/rapm-2024-106130. Online ahead of print. PMID 39740957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2019 and February 2023, a total of 110 eligible patients were randomized and 55 were assigned to each treatment group, 1% Chloroprocaine or 0.75% Bupivacaine. Study was paused from March 2020 to September 2020 due to the pandemic and was also paused December 2020 because the surgery center was closed and the pharmacy was unable to obtain the necessary medications from the manufacturer.
Period: Overall Study
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
Started | 55 | 55
Completed | 54 | 51
Not Completed | 1 | 4
Not completed — Inability to place a spinal anesthesia due to the patients' anatomy | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 50.5 [45.0 to 58.0] | 48.0 [36.0 to 59.0] | 49.3 [40.6 to 58.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 35 | 30 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54 | 51 | 105
American Society of Anesthesiologists Physical Status (ASA-PS) Classification [Count of Participants; unit: Participants] — Patients physical status at baseline was recorded using the American Society of Anesthesiologists Physical Status (ASA-PS) classification. Healthy patients with no significant systemic disease were classified as Class I. Patients with mild systemic disease that did not significantly limit daily activities were classified as Class II. Patients with severe systemic disease that limited daily activities were classified as Class III. Results have been summarized by study arm.
  Participants
    Class I | 0 | 4 | 4
    Class II | 40 | 37 | 77
    Class III | 14 | 10 | 24
Body Mass Index (BMI) [Mean (Inter-Quartile Range); unit: kg/m^2] — BMI data was collected at baseline and summarized by study arm.
  kg/m^2 | 29.1 [24.4 to 31.7] | 28.1 [24.4 to 32.3] | 28.6 [24.4 to 32.0]
Surgical Procedure [Count of Participants; unit: Participants] — The type of anorectal procedure performed is summarized by study arm.
  Participants
    Ablation | 24 | 22 | 46
    Anal Fissurectomy | 8 | 5 | 13
    Debridement | 6 | 8 | 14
    Exam Under Anesthesia | 8 | 3 | 11
    Hemorrhoidectomy | 7 | 12 | 19
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time
Description: For this study Recovery time was defined as the time (in minutes) to return of both motor and sensory function, postoperatively. The return of motor function was tested by demonstrating mobility in both lower extremities including hips, knees, and lower legs using the Bromage scale. The return of sensory function was assessed using light touch and/or pinprick techniques on the dermatomes corresponding with the T8-S2 spinal cord segments. The duration in minutes when both sensory and motor function were re-established was documented and results were summarized by study arm using basic descriptive statistics. In this study it is hypothesized that use of 1% Chloroprocaine spinal anesthesia will reduce recovery times of patients undergoing anorectal procedures as compared to 0.75% bupivacaine spinal.
Time Frame: On post-operative day 1 (POD1), approximately every 15 minutes up to 24 hours
Measure: Mean (Standard Error); unit: minutes
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
Number analyzed (Participants) | 54 | 51
minutes | 134.1 (8.6) | 161.9 (10.3)

2. Primary Outcome: Discharge Time
Description: For this study discharge time is defined as the time (in minutes) when the patient is "fit to discharge" from the Postoperative Care Unit (PACU). At the institution where this study took place "fit to discharge" was defined as the ability to void and the ability to ambulate unassisted for at least 10 feet. The duration of time when a patient was able to do both was documented. Results were summarized by study arm using basic descriptive statistics. It is hypothesized that the use of 1% Chloroprocaine spinal anesthesia will result in a clinically significant 30% reduction in discharge times of patients as compared to 0.75% bupivacaine spinal.
Time Frame: On post-operative day 1 (POD1), up to 24 hours
Measure: Mean (Standard Error); unit: minutes
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
Number analyzed (Participants) | 54 | 51
minutes | 191.4 (6.6) | 230.9 (9.4)

3. Secondary Outcome: Evidence of Hypotension
Description: Evidence of hypotension will be documented if systolic blood pressure (SBP) drops more than 20mmHg from baseline following spinal anesthesia. Hypotension is a common side effect of spinal anesthesia (SA). The number of participants with evidence of hypotension will be summarized by study arm.
Time Frame: On day of procedure, 0-5 minutes following administration of spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
Number analyzed (Participants) | 54 | 51
Participants | 0 | 0

4. Secondary Outcome: Evidence of Transient Neurological Symptoms (TNS)
Description: The number of participants demonstrating TNS approximately 24 hours following the procedure will be assessed. TNS will be defined as back pain or dysesthesia that radiated to the buttocks, thighs, hips, or calves and began within the first 24 hours after surgery. Localized pain or tenderness at the injection site or lower back without radiation will not be considered TNS. TNS is clinically important as it causes patient pain and discomfort and, in severe cases, may delay discharge or cause readmission. Symptoms will be summarized and reported by study arm.
Time Frame: On post-op day 2, approximately 24 hours post operation
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
Number analyzed (Participants) | 54 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 hours following procedure
Arm/Group | 1% Chloroprocaine (PF) | 0.75% Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03324984/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03324984/ICF_001.pdf